CLINICAL TRIAL: NCT02584036
Title: Project IMPACT Immunizations (IMProving America's Communities Together)
Status: Completed | Type: Observational
Sponsor: American Pharmacists Association Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 015
Record Dates: First submitted 2015-10-20; First posted 2015-10-22 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Influenza
Keywords: influenza; vaccine; public health; preventable disease; vaccine history; point-of-care
MeSH Terms: conditions — Influenza, Human | interventions — Proto-Oncogene Proteins c-met; Patient Education as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Receiving Influenza Vaccine: Patients who receive an influenza vaccine at a participating pharmacy site will be eligible to: a) receive a vaccination forecast review, b) be evaluated for unmet vaccination needs, c) receive patient education, and d) have vaccination needs met.
  Interventions: Biological: Vaccine administration by a pharmacist; Behavioral: Unmet vaccination needs identified and met; Behavioral: Vaccination forecast review and patient education

INTERVENTIONS:
Biological: Vaccine administration by a pharmacist — Administration, number and types, of vaccine(s) by a pharmacist
Behavioral: Unmet vaccination needs identified and met — Identification of unmet vaccination needs and having those needs met
Behavioral: Vaccination forecast review and patient education — Pharmacist review of the vaccination forecast and patient education on his/her vaccine needs

SUMMARY:
The primary objective of this study is to evaluate how implementing an innovative care model that provides the pharmacist access to a patient's vaccine history at the point-of-care impacts the pharmacist's ability to identify unmet vaccination needs and increase vaccination rates for routinely recommended adult vaccinations.

DETAILED DESCRIPTION:
This is a multi-site, observational study investigating the impact of implementing an innovative care model on the pharmacist's ability to identify unmet vaccination needs and increase vaccination rates for routinely recommended adult vaccinations. The innovative care model enables the pharmacist to utilize a bi-directional IIS to assess patients' vaccination histories, identify unmet vaccination needs, and document the care provided. Data will be collected in the bi-directional IIS. Aggregate de-identified data will be reported to the researchers at the midpoint and conclusion of the study. The project duration has been established to allow sufficient time for each pharmacy to implement the innovative care model and monitor each pharmacy for a 6-month study period. The American Pharmacists Association (APhA) Foundation has an a priori intent to publish the project results.

ELIGIBILITY:
Inclusion Criteria:

* Individuals eligible to be enrolled in the study include any person at least 18 years of age receiving an influenza vaccination from a participating pharmacy site.

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients receiving an influenza vaccine
Sampling Method: Non-Probability Sample
Enrollment: 1080 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number and types of vaccines administered | Change from baseline rates at 6 months
Number of unmet vaccination needs identified and met | through study completion, an average of 6 months
Number of times the pharmacist reviewed the vaccination forecast and educated the patient on his/her vaccine needs | through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin M Bluml, BPharm, Principal Investigator — American Pharmacists Association
Locations (8):
- United States (8):
  - Quality Food Centers #101, Belfair, Washington
  - Cheney-Owl Pharmacy, Cheney, Washington
  - Kirk's Pharmacy, Eatonville, Washington
  - Quality Food Centers #851, Edmonds, Washington
  - Lopez Island Pharmacy, Lopez Island, Washington
  - Kelley-Ross Pharmacy, Seattle, Washington
  - ReliantRx, Spokane, Washington
  - Tieton Village Drug, Yakima, Washington